CLINICAL TRIAL: NCT02130713
Title: Chronic Bacterial Prostatitis: Efficacy of Short-lasting Antibiotic Therapy With Prulifloxacin (Unidrox®) in Association With Saw Palmetto Extract, Lactobacillus Sporogens and Arbutin (Lactorepens®)
Brief Title: Treatment of Chronic Bacterial Prostatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Ettore De Berardinis, Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1611380961111745
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Bacterial Prostatitis
MeSH Terms: conditions — Prostatitis | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A, antibiotics (Active Comparator): Prulifloxacin 600 mg
  Interventions: Drug: Third generation fluoroquinolone
- Group B, antibiotics plus nutraceuticals (Active Comparator): Prulifoxacin plus Serenoa repens 320 mg, Lactobacillus Sporogens 200 mg, Arbutin 100 mg
  Interventions: Dietary Supplement: Nutritional supplement + third generation fluoroquinolone

INTERVENTIONS:
Drug: Third generation fluoroquinolone — Prulifloxacin 600 mg
  Arms: Group A, antibiotics
Dietary Supplement: Nutritional supplement + third generation fluoroquinolone — Serenoa repens 320 mg, Lactobacillus Sporogens 200 mg, Arbutin 100 mg and prulifloxacin 600 mg
  Arms: Group B, antibiotics plus nutraceuticals

SUMMARY:
Background - bacterial prostatitis (BP) is a common condition accounting responsible for about 5-10% of all prostatitis cases; chronic bacterial prostatitis (CBP) classified as type II, are less common but is a condition that significantly hampers the quality of life, (QoL) because not only is it a physical condition but also a psychological distress. Commonly patients are treated with antibiotics alone, and in particular fluoroquinolones are suggested by the European Urology guidelines. This approach, although recommended, may not be enough. Thus, a multimodal approach to the prolonged antibiotic therapy may be helpful.

Methods - 210 patients affected by chronic bacterial prostatitis were enrolled in the study. All patients were positive to Meares-Stamey test and symptoms duration was > 3 months. The purpose of the study was to evaluate the efficacy of a long lasting therapy with a fluoroquinolone in association with a nutraceutical supplement (prulifloxacin 600 mg for 21 days and an association of Serenoa repens 320 mg, Lactobacillus Sporogens 200 mg, Arbutin 100 mg for 30 days). Patients were randomized in two groups (A and B) receiving respectively antibiotic alone and an association of antibiotic plus supplement.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by chronic bacterial prostatitis
* positivity to the Meares-Stamey test
* symptoms duration > 3 months (dysuria, pelvic pain and/or discomfort)

Exclusion Criteria:

* positivity to Chlamydia trachomatis, Ureaplasma urealiticum, Mycoplasma, Neisseria gonorrhoeae, herpes simplex viruses (HSV 1/2) and human papillomavirus (HPV)
* age less than 18 years
* history of neurological disease, urinary stones or cancer
* allergy to fluoroquinolones
* refusal to sign the informed consent
* incomplete follow-up time.

Ages: 19 Years to 54 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Meares-Stamey evaluation | up to 6 months
  The Meares-Stamey test, also known as 4-glass test, is the standard method of assessing inflammation and presence of bacteria in the lower urinary tract of men presenting CBP. The test has been performed on each patient before and after the therapy. The Meares-Stamey evaluation allows the collection of four samples: first voided urine (VB1) that represents urethra, mid-stream urine (VB2) that represents bladder, expressed prostatic secretion (EPS) and post-prostatic massage urine (VB3) that represent the prostate. It is considered positive when we have urophathogen colony-forming units (CFU)/mL ≥103.

SECONDARY OUTCOMES:
NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) | up to 6 months
  The NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) is a questionnaire with 13 questions developed to evaluate symptoms and quality of life in men with chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). Every question has a score differing by the answer, and the questionnaire has a total score ranging from 0 to 43. The score is divided by three subscales: pain (score range 0-21), urinary symptoms (score range 0-10) and quality of life (QoL) (score range 0-12). The sum of all single scores is the total score. The reason every item has a different maximum score is because they have a different potential. NIH-CPSI characteristics are: good reliability, validity, and responsiveness to change. It has been used in many large-scale trials regarding CP/CPPS as the primary outcome variable [14].

CONTACTS AND LOCATIONS:
Overall Officials: Ettore De Berardinis, Professor, Study Director — Policlinico Umberto I - Department of Gynecological-Obstetrics Sciences and Urological Sciences
Locations (1):
- policlinico Umberto I - Department of Gynecological-Obstetrics Sciences and Urological Sciences, Roma, Roma, Italy

REFERENCES:
- [Derived] Busetto GM, Giovannone R, Ferro M, Tricarico S, Del Giudice F, Matei DV, De Cobelli O, Gentile V, De Berardinis E. Chronic bacterial prostatitis: efficacy of short-lasting antibiotic therapy with prulifloxacin (Unidrox(R)) in association with saw palmetto extract, lactobacillus sporogens and arbutin (Lactorepens(R)). BMC Urol. 2014 Jul 19;14:53. doi: 10.1186/1471-2490-14-53. PMID 25038794